CLINICAL TRIAL: NCT00456872
Title: A Contrast of Buffered Vs. Unbuffered Lidocaine in Bone Marrow Biopsies
Brief Title: Contrast of Buffered Vs. Unbuffered Lidocaine in Bone Marrow Biopsies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0457
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Pain
Keywords: Pain during injection of the pre-procedure anesthetic
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- buffered lidocaine (Experimental): Sodium bicarbonate is a buffering additive that decreases the pH of the solution allowing for decrease in pain upon filtration.
  Interventions: Drug: lidocaine
- unbuffered lidocaine (Experimental): lidocaine is injected without sodium bicarbonate added
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: lidocaine
  Other Names: Xylocaine; lignocaine

SUMMARY:
Oncology patients require numerous invasive procedures throughout their disease process including bone marrow biopsies (BMB). BMB.s are performed by a significant number of health care providers. One of the biggest concerns for health care providers is to improve patient comfort. The goal of this study was to reduce pain during BMBs.

Specific aims of the study were to determine if there is a difference in patients' perceived pain during injection of the pre-procedure anesthetic when buffered versus unbuffered lidocaine is administered to patient's receiving bone marrow biopsies.

A double blind, experimental crossover design was used to examine the difference in pain levels when using buffered versus unbuffered lidocaine prior to the bilateral bone marrow biopsy procedure. Based on a power analysis for a paired t-test, a convenience sample of 48 patients was enrolled into the study. Patients served as their own control. The site of first biopsy, and which lidocaine solution was administered first, were randomized. A 100mm visual analogue scale (VAS) was used to measure pain.

All data has been collected, are currently under analysis, and results will be completed in August 2006. Differences in groups will be examined using a paired t-test. A demographic questionnaire was used to gather select demographic variables. Correlative studies will be done to examine the relationship between the patient's perceived pain scores and several exploratory variables. Results of this study may change the current type of anesthetic used pre-BMBs thus improving patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Any newly diagnosed patient at the Arthur G. James Cancer Hospital and Richard J. Solove Research Institute whose Hematologist or Oncologist has ordered them to undergo a bilateral bone marrow biopsy for diagnostic and /or treatment purposes.
* 18 years of age or older.

Exclusion Criteria:

* Pregnant or Lactating women.
* Patients with allergies to local anesthetics.
* Patients requiring a unilateral bone marrow biopsy.
* Patients that cannot lie flat in either the supine or prone position.
* Patients that have used any of the following: narcotics, non-narcotic analgesia or an anti-anxiolytic medication on the same calendar day as the scheduled procedure. These medications will not be given to the participant at any time before or during the procedure.
* Patients on long-acting narcotic medication.
* Patients with neuropathy in the posterior iliac crest area
* Patients with a platelet count less than 20,000.
* Patients who are cognitively impaired or unable to self-report pain using the VAS.
* Patients with known bone metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-12; Primary Completion 2006-05 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Difference in patients perceived pain during injection of the pre-procedure anesthetic | Up to 24 months
  Determine difference in patients perceived pain during injection of pre-procedure anesthetic when buffered versus unbuffered lidocaine is administered.

SECONDARY OUTCOMES:
Change in pain level over time after anesthetic is administered. | Up to 24 months
  Determine if pain levels change over time after anesthetic is administered.
Investigate relationships between patients perceived pain scores and variables. | Up to 24 months
  Variables include gender, ethnicity, stage and extent of disease, body mass index, history of pain tolerance, and perceived emotional support.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Hollar-Ruegg, MS, RN, CNP, AOCN, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University James Cancer Hospital, Columbus, Ohio, United States

REFERENCES:
- [Result] Ruegg TA, Curran CR, Lamb T. Use of buffered lidocaine in bone marrow biopsies: a randomized, controlled trial. Oncol Nurs Forum. 2009 Jan;36(1):52-60. doi: 10.1188/09.ONF.52-60. PMID 19136338
- See also: Jamesline — http://cancer.osu.edu